CLINICAL TRIAL: NCT04230018
Title: A Study Comparing the Gene Profiles of Primary and Heterogeneous Metastases of Colorectal Cancer
Brief Title: The Gene Profiles of Primary and Heterogeneous Metastases of Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Dean, Chief Physician, headof Gastroenterology, Professor#Principal Investigator, Clinical Professor, Sun Yat-sen University
Other Study IDs: Gene primary versus metastases
Record Dates: First submitted 2019-10-28; First posted 2020-01-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC; primary focus; metastasis; heterogeneous metastasis; gene
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- primary and metastasis lesion: tissue of colorectal cancer primary lesion and tissue of colorectal cancer metastasis were obtained

SUMMARY:
The incidence and mortality of colorectal cancer in China's cancer disease spectrum is on the rise, and it is a common malignant tumor that harms the health of Chinese residents.In patients with synchronous metastatic colorectal cancer, RAS status is highly consistent in primary focus and metastasis, so NCCN guidelines recommend RAS testing of primary or metastatic tissue is feasible .However, there are also some reports that the difference of RAS status between primary and metastatic lesions was up to 22%.In additiont,there are few studies on whether the gene profile of the metastatic lesion is the same as that of the primary lesion in patients with postoperative heterogeneous metastasis in patients with stage III colorectal cancer.

DETAILED DESCRIPTION:
The incidence and mortality of colorectal cancer in China's cancer disease spectrum is on the rise, and it is a common malignant tumor that harms the health of Chinese residents. Now NCCN guidelines recommend targeted drugs for the treatment of metastatic colorectal cancer mainly including cetuximab and panizumab whic targeting EGFR , as well as the bevacizumab and arber regofini, etc which targeing anti-angiogenic.Cetuximab and panizumab are only effective in patients with RAS wild type.

Previous studies have shown that In patients with synchronous metastatic colorectal cancer, RAS status is highly consistent in primary focus and metastasis, so NCCN guidelines recommend RAS testing of primary or metastatic tissue is feasible .However, there are also some reports that the difference of RAS status between primary and metastatic lesions was up to 22%.In additiont,there are few studies on whether the gene profile of the metastatic lesion is the same as that of the primary lesion in patients with postoperative heterogeneous metastasis in patients with stage III colorectal cancer.

Therefore, it has important clinical significance to compare the difference of gene profile between metastatic lesion and primary lesion in patients with postoperative metastasis of stage III colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 75 years old, both men and women;
2. Patients must have histologically confirmed metastatic colorectal adenocarcinoma and metastases can be punctured by interventional evaluation;
3. ECOG: 0 to 2;
4. Expected survival ≥ 12 weeks;
5. Absolute neutrophil count (ANC) ≥ 1.5 × 109 /L; Hemoglobin ≥ 8g / dL; Platelets ≥100×109/L;(According to the normal value of the clinical trial center)
6. Prothrombin time (PT) < 1.5 times the upper normal limit and thrombin time (APTT) < 1.5 times the upper normal limit;
7. Informed consent has been signed.

Exclusion Criteria:

1. Patients had surgery within three weeks will be excluded.
2. Patients have known or suspected brain metastases will be excluded.
3. Pregnant or nursing women will be excluded.
4. Patients with severe uncontrolled systemic disease, such as severe active infection, will be excluded.
5. Patients had other malignancies in the past 5 years will be excluded, except cervical carcinoma in situ or basal cell carcinoma of the skin.
6. Patients who were unable to complete the study or sign valid informed consent for medical, social or psychological reasons, which will be determined by researcher, will be excluded.
7. Organ transplant recipients who need immunosuppressive therapy will be excluded.
8. People have been known to be infected with immunodeficiency virus (HIV) or have been known to be serologically positive for HIV will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with postoperative heterochronous metastasis,who has histologically confirmed metastatic colorectal adenocarcinoma and metastases could be punctured by interventional evaluation.In addittion,patients' blood ctDNA and tissues can be used to detect genetic mutations.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-12-28 (Actual); Primary Completion 2021-12-27 (Estimated); Study Completion 2021-12-27 (Estimated)

PRIMARY OUTCOMES:
Mutation Consistency of metastatic and primary sites of colorectal cancer patients with postoperative metastasis | through study completion, an average of 2 years.
  We do NGS sequencing of both the primary and metastatic tissue sample of the CRC patients. The gene mutation data will be analysis, and the percentage of same and different mutation of the samples will be compared.

SECONDARY OUTCOMES:
Mutation Consistency of tissue and blood sample | through study completion, an average of 2 years.
  The gene mutation data will be analysis, and the percentage of same and different mutation of the samples will be reported. The consistency between the gene mutation of ctDNA test in blood and the gene mutation of tissue test is analyzed to determine whether the blood ctDNA test could replace the tissue gene test

OTHER OUTCOMES:
prediction accuracy of survival rate | through study completion, an average of 2 years.
  We will use the gene mutation data and follow-up data of the patients to construct a prediction model, and the accuracy of model to anticipating the 2-year survival rate of patients will be analyzed. To analyze the relationship between different gene mutations and patients' recurrence and prognosis, and to clarify the prognostic role of new mutations in heterogeneous metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siyar Ekinci A, Demirci U, Cakmak Oksuzoglu B, Ozturk A, Esbah O, Ozatli T, Celik B, Budakoglu B, Turker I, Bal O, Turan N. KRAS discordance between primary and metastatic tumor in patients with metastatic colorectal carcinoma. J BUON. 2015 Jan-Feb;20(1):128-35. PMID 25778307